CLINICAL TRIAL: NCT06107023
Title: Investigation of the Effect of Action Observation Training With 3D Virtual Reality on Upper Extremity Functions in Patients With Multiple Sclerosis With Attacks
Brief Title: Action Observation Training With 3D Virtual Reality in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuba Kaya Benli, lecturery, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-TKB-001
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; motor learning; action observation training; virtual reality; upper extremity function
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): action observation and upper extremity activities
  Interventions: Behavioral: Action observation training
- Control Group (Sham Comparator): sham action observation and upper extremity activities
  Interventions: Behavioral: sham action observation training

INTERVENTIONS:
Behavioral: Action observation training — 6 weeks, three days a week.
  Arms: Intervention Group
Behavioral: sham action observation training — 6 weeks, three days a week.
  Arms: Control Group

SUMMARY:
Multiple sclerosis is a chronic, autoimmune and inflammatory disease of the Central Nervous System characterized by neuronal demyelination and axonal degeneration. Upper extremity problems are present in MS patients from an early stage, affecting the performance of the individual and leading to a decrease in activity of daily living ability in proportion to the extent of the problem. Action Observation Training is currently being examined as one of the methods used for the improvement of motor disorders and has been shown in the literature to be effective on different functions in neurological diseases.

The aim of this study was to investigate the effects of action observation training with 3D virtual reality on upper extremity functions, fatigue, cognitive functions, activities of daily living and quality of life in MS patients.

Hypothesis 1: Action observation training with 3D virtual reality has an effect on upper extremity functions in MS patients.

Hypothesis 2: Action observation training with 3D virtual reality has an effect on cognitive function in MS patients.

Hypothesis 3: Action observation training with 3D virtual reality has an effect on fatigue in MS patients.

Hypothesis 4: Action observation training with 3D virtual reality has an effect on activities of daily living in MS patients.

Hypothesis 5: Action observation training with 3D virtual reality has an effect on quality of life in MS patients.

DETAILED DESCRIPTION:
The training will involve watching 3D videos of upper limb functions in VR and then repeating the functions by the participants. The AOT group will watch video sequences involving upper limb functions, while the control group will watch landscape videos that are not likely to elicit activity in motor or ANS areas.

In our study, 3D videos of upper limb functions will be recorded with a 360° camera and will be shown to individuals through the VR system from the primary person's perspective.

ELIGIBILITY:
Inclusion Criteria:

* < 2 years MS diagnosis according to McDonald criteria
* between 3.5 and 6 the EDSS
* Nine Hole Peg Test > 30s for at least one upper extremity
* no change in medication in the last 6 months
* having MS disease with ongoing attacks
* >2 Modified Ashworth Scale in the upper extremities
* MOCA>25

Exclusion Criteria:

* diagnosed with neurological (except MS), cardiopulmonary, metabolic or musculoskeletal disease that would prevent treatment and evaluation
* receiving botulinum toxin treatment in the last 6 months
* visual impairment uncorrected by optical devices
* inability to adapt to treatment based on 3D immersive virtual reality (e.g. with cognitive impairment, communication problems, psychological problems or vestibular system problems)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | baseline and 6th week
  upper extremity function assessment
nine hole peg test | baseline and 6th week
  upper extremity function assessment
hand dynamometer | baseline and 6th week
  grip strength assessment

SECONDARY OUTCOMES:
Fatigue severity scale | baseline and 6th week
  fatigue assessment
Paced Auditory Serial Addition Test | baseline and 6th week
  Cognitive assessment
The Arm Function in Multiple Sclerosis Questionnaire | baseline and 6th week
  activities of daily living assessment
Multiple Sclerosis Quality of Life-54 | baseline and 6th week
  quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Kaya Benli, MSc, Principal Investigator — Abant Izzet Baysal University; Yeşim Bakar, Prof. Dr., Study Director — Izmir Bakircay University; Şule Aydın Türkoğlu, Assoc. Prof., Study Chair — Abant Izzet Baysal University; Enes Tayyip Benli, MSc, Study Chair — Abant Izzet Baysal University
Locations (1):
- Izzet Baysal University, Bolu, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bunday KL, Lemon RN, Kilner JM, Davare M, Orban GA. Grasp-specific motor resonance is influenced by the visibility of the observed actor. Cortex. 2016 Nov;84:43-54. doi: 10.1016/j.cortex.2016.09.002. Epub 2016 Sep 11. PMID 27697663
- [Background] Choi JW, Kim BH, Huh S, Jo S. Observing Actions Through Immersive Virtual Reality Enhances Motor Imagery Training. IEEE Trans Neural Syst Rehabil Eng. 2020 Jul;28(7):1614-1622. doi: 10.1109/TNSRE.2020.2998123. PMID 32634098
- [Background] Rocca MA, Meani A, Fumagalli S, Pagani E, Gatti R, Martinelli-Boneschi F, Esposito F, Preziosa P, Cordani C, Comi G, Filippi M. Functional and structural plasticity following action observation training in multiple sclerosis. Mult Scler. 2019 Oct;25(11):1472-1487. doi: 10.1177/1352458518792771. Epub 2018 Aug 7. PMID 30084706
- [Background] Sollfrank T, Hart D, Goodsell R, Foster J, Tan T. 3D visualization of movements can amplify motor cortex activation during subsequent motor imagery. Front Hum Neurosci. 2015 Aug 20;9:463. doi: 10.3389/fnhum.2015.00463. eCollection 2015. PMID 26347642
- [Background] Yoshimura M, Kurumadani H, Hirata J, Osaka H, Senoo K, Date S, Ueda A, Ishii Y, Kinoshita S, Hanayama K, Sunagawa T. Virtual reality-based action observation facilitates the acquisition of body-powered prosthetic control skills. J Neuroeng Rehabil. 2020 Aug 20;17(1):113. doi: 10.1186/s12984-020-00743-w. PMID 32819412
- [Background] Yu JA, Park J. The effect of first-person perspective action observation training on upper extremity function and activity of daily living of chronic stroke patients. Brain Behav. 2022 May;12(5):e2565. doi: 10.1002/brb3.2565. Epub 2022 Apr 10. PMID 35398981